CLINICAL TRIAL: NCT06917248
Title: Evaluation of Clinical Effectiveness and Safety of Locaste 8F Guiding Catheter in Neurovascular Interventional Surgery
Status: Completed | Type: Observational
Sponsor: Keuro MedTech (Industry)
Responsible Party: Sponsor
Other Study IDs: CIP-PICA-RWD
Record Dates: First submitted 2025-03-21; First posted 2025-04-08 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Stroke; Hemorrhagic Strokes
Keywords: Locaste; Long sheath; Guiding catheter
MeSH Terms: conditions — Stroke; Hemorrhagic Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Locaste 8F Guiding Catheter in Neurovascular interventional surgery: Patients with Locaste 8F Guiding Catheter used in the neurovascular interventional surgery and the surgery video of the Locaste 8F Guiding Catheter available are recruited in this study.

SUMMARY:
The Locaste 8F Delivery Catheter by Kai MedTech has been launched in China since 2022 and has been widely used clinically. It won the government tendering in many provinces in China in early 2024. As a guiding and access device, the investigational device is used in interventional surgeries. The clinical investigation plans to conduct a non-interventional post-marketing real-world study to evaluate the safety and effectiveness of the product in clinical use. The investigator shall use the Locaste 8F Guiding Catheter according to his own surgery plan and the instruction for use (IFU) of this device. The large-bore guiding catheters (also called as long guiding sheath) by global manufacturers are generally used. Locaste 8F Guiding Catheter is marketed in China and widely accepted in clinical application. By collecting data in the real-world clinical routine treatment, the effectiveness and the safety of Locaste 8F Guiding Catheter is evaluated to provide data support of further global use of this device.

DETAILED DESCRIPTION:
This clinical investigation is a single-arm, retrospective, multicenter clinical study of a medical device marketed in China. Patients with Locaste 8F Guiding Catheter used in the neurovascular interventional surgery and the surgery video of the Locaste 8F Guiding Catheter available are recruited in this study. The data on the surgery day and follow-up data within 24 hours after surgery are collected retrospectively.

This clinical investigation will be performed in accordance with the Declaration of Helsinki [5] and the applicable parts of ISO 14155：2020 Clinical investigation of medical devices for human subjects - Good clinical practice made by International Organization for Standardization except for section 5.8 informed consent and other non-relevant aspects for retrospective study. The ethic approval was achieved with the exemption of informed consent according to the local China regulations "The Guidelines for the Establishment of Ethical Review Committees for Clinical Research Involving Humans", article 5 Exemption of Informed consent.

Since this clinical investigation is a non-interventional post-market study with the intended use of the investigational device in China, this study does not apply to the scope of pre-market clinical investigation for medical device approval defined in the Medical Device Good Clinical Practice (2022) issued by the China NMPA . Thus, this clinical investigation only refers to the applicable part of the Medical Device Good Clinical Practice (2022) issued by the China NMPA.

Given the fact that this clinical investigation is a retrospective study, any serious adverse event (SAE) should have been reported according to the regulation Procedure for Monitoring and Re-evaluation of Medical Device Adverse Event (2018). No serious adverse events in this study shall be reported again. In case of any underreporting, the investigator shall report the serious adverse events according to the Procedure for Monitoring and Re-evaluation of Medical Device Adverse Event (2018).

The intended use of the investigational device approved in China is that "The device is indicated for the introduction of interventional devices into the peripheral, coronary, and neuro vasculature". The subject cohort in this clinical investigation is covered by the device use scope.

ELIGIBILITY:
Inclusion Criteria:

* Age of 18 years or older;
* Undertaken a neurovascular surgery procedure including Locaste 8F Guiding Catheter;
* Available images of Locaste 8F Guiding Catheter in the neurovascular surgery;

Exclusion Criteria:

* Disorders of vascular fragility (e.g. Ehlers-Danlos syndrome)
* Prior vascular dissection or injury to vessels to be catheterized

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undertaken a neurovascular intervention surgery procedure including Locaste 8F Guiding Catheter in a reverse chronological order earlier than the date of the ethic approval.
Sampling Method: Non-Probability Sample
Enrollment: 113 (Actual)
Dates: Start 2024-05-21 (Actual); Primary Completion 2024-10-07 (Actual); Study Completion 2024-10-07 (Actual)

PRIMARY OUTCOMES:
Device Success Rate | Day 0 （During surgery）
  Definition：Number of Patients with Device Success / Number of Recruited Patients * 100% Device Success： Use 5-Point Likert Scale to evaluate the navigability of device to the targeted vessel position.
  1. Unsatisfactory；
  2. Unacceptable；
  3. Adequate；
  4. Good;
  5. Excellent； Device success is defined as the score ≥3.

SECONDARY OUTCOMES:
Ability to deliver other interventional devices | Day 0（During surgery）
  Definition：the incidence of score ≥3: Ability to deliver other interventional devices is defined the satisfactory rate of the ability to deliver other interventional devices. Use 5-Point Likert Scale to evaluate the ability to deliver other interventional devices.
  1. Unsatisfactory；
  2. Unacceptable；
  3. Adequate；
  4. Good；
  5. Excellent；
Visibility under X-ray | Day 0（During surgery）
  Definition：Visibility under X-ray: the incidence of score ≥3； Visibility under X-ray is defined as the satisfactory rate of the visibility under X-ray. Use 5-Point Likert Scale to evaluate the Visibility under X-ray.
  1. Unsatisfactory；
  2. Unacceptable；
  3. Adequate；
  4. Good；
  5. Excellent；
Ability to support other interventional devices | Day 0（During surgery）
  The incidence to achieve satisfactory support of other interventional devices.
Device Deficiency | Day 0 (During surgery)
  For all the subjects who have completed the surgery, no defects of the investigational device were found. One patient did not complete the surgery and no defects of the investigational device were found during the use.
Adverse Event (AE) | Day 0(during surgery) or Day 1 (within 24 hours after the surgery)
  For all the subjects who have completed the surgery, no adverse events were found. One patient did not complete the surgery and no adverse events were found during the use.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Xinxiang City Central Hospital, Xinxiang, Henan
  - Zhumadian City Central Hospital, Zhumadian, Henan

IPD SHARING:
Plan to Share IPD: Undecided